CLINICAL TRIAL: NCT01170481
Title: Retinal Nerve Fibre Layer in Uveitic Secondary Glaucoma
Brief Title: Assessment of Retinal Nerve Fibre Layer by Optical Coherence Tomography in Uveitis Patients With Papilloedema
Status: Completed | Type: Observational
Sponsor: St. Franziskus Hospital (Other)
Responsible Party: Principal Investigator, Carsten Heinz, Head of Department, St. Franziskus Hospital
Other Study IDs: 2008-128-f-S
Record Dates: First submitted 2010-07-21; First posted 2010-07-27 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Uveitis; Glaucoma
Keywords: anterior and intermediate uveitis; papilloedema
MeSH Terms: conditions — Uveitis; Glaucoma; Uveitis, Intermediate; Papilledema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- papilloedema without glaucoma
- papilloedema with glaucoma
- glaucoma without papilloedema

SUMMARY:
Assessment of optic disc morphology can be difficult in patients with uveitis and papilloedema. Therefore different optical coherence tomography (OCT) and laser scanning techniques may help to detect damage to the retinal nerve fibre layer.

ELIGIBILITY:
Inclusion Criteria:

* anterior or intermediate uveitis
* papilloedema
* glaucoma

Exclusion Criteria:

* dense cataract
* dense vitreous opacification
* circular posterior synechiae

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with anterior or intermediate uveitis and papillooedema in fluoreszein angiography.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Alterations of retinal nerve fibre layer by optical coherence tomography | once at study entry
  Baseline comparision of retinal nerve fibre layer thickness in patients with uveitis and with or without papilloedema at study entry. No follow-up examination scheduled

CONTACTS AND LOCATIONS:
Overall Officials: Arnd Heiligenhaus, MD, Study Chair — Department at St. Franziskus Hospital
Locations (1):
- Department of Ophthalmology at St.-Franziskus Hospital, Münster, Germany

REFERENCES:
- [Derived] Heinz C, Kogelboom K, Heiligenhaus A. Influence of optic disc leakage on objective optic nerve head assessment in patients with uveitis. Graefes Arch Clin Exp Ophthalmol. 2016 Feb;254(2):361-4. doi: 10.1007/s00417-015-3218-5. Epub 2015 Nov 18. PMID 26582161
- See also: Related Info — http://www.uveitis-zentrum.de